CLINICAL TRIAL: NCT00392431
Title: Continuous Versus Episodic Prophylactic Treatment With Oral Amiodarone for the Prevention of Permanent Atrial Fibrillation: a Randomized Study on Morbidity and Quality of Life
Brief Title: Continuous Versus Episodic Amiodarone Treatment for the Prevention of Permanent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Netherlands Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000B133
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2007-03-22 (Estimated); Status verified 2007-03

CONDITIONS: Persistant Atrial Fibrillation
MeSH Terms: interventions — Amiodarone

INTERVENTIONS:
Drug: amiodarone

SUMMARY:
Our hypothesis is that episodic amiodarone treatment (i.e. amiodarone treatment 1 month prior until 1 month after cardioversion) is associated with a lower morbidity and a higher quality of life compared to continuous prophylactic amiodarone treatment while atrial fibrillation is still effectively suppressed. The latter means that at the end of the study permanent atrial fibrillation is prevented in comparable percentage of patients (70%) in both treatment strategies. However, this will be accomplished at the cost of a higher number of electrical cardioversions (2-3) in the episodic treatment group compared to the continuous treatment group.

DETAILED DESCRIPTION:
Primary objective

To determine differences in adverse event rates between patients with persistent atrial fibrillation who are randomized to episodic amiodarone treatment (EAT) strategy and patients who are randomized to continuous amiodarone treatment (CAT) strategy, while atrial fibrillation is still effectively suppressed.

Adverse events can be related to:

1. amiodarone use
2. atrial fibrillation itself or underlying heart disease.

Secondary objective

To determine differences in quality of life between patients with persistent atrial fibrillation who are randomized to the EAT strategy and patients who are randomized to the CAT strategy.

ELIGIBILITY:
Inclusion criteria:

1. Symptomatic persistent atrial fibrillation for at least 48 hours- 1 year (present episode).
2. Older than 18 years of age.
3. Ventricular rate during AF > 75 beats per minute, documented on rest-ECG without rate control.
4. At least two weeks of oral anticoagulation therapy before screening.
5. Written informed consent.

Exclusion criteria:

1. Contra indications for amiodarone (severe chronic obstructive pulmonary disease or QTc > 440ms).
2. History of relapse of AF during adequate amiodarone treatment (i.e. adequate amiodarone and desethylamiodarone plasma levels).
3. Concomitant treatment with class I or III antiarrhythmic drugs. Amiodarone should not have been used during the last 3 months.
4. Other (non) cardiac QT prolonging drugs (if not possible to discontinue).
5. First episode of persistent atrial fibrillation.
6. More than three relapses of persistent atrial fibrillation necessitating electrical cardioversion during the last three years.
7. Known sick sinus syndrome.
8. History of second or third degree AV conduction disturbances.
9. Intraventricular conduction disturbances (QRS> 140ms).
10. Pacemaker treatment.
11. Hemodynamically significant valvular disease.
12. Patients with heart failure with symptoms according to NYHA class III or IV.
13. Unstable angina pectoris.
14. Recent myocardial infarction (< 3 months).
15. PTCA, CABG, other cardiac surgery or major non-cardiac surgery within the last three months.
16. History of hyperthyroidism or hypothyroidism.
17. Serious pulmonary, hepatic, haematological, metabolic, renal, gastrointestinal, CNS or psychiatric disease.
18. Pregnant and non-pregnant women who are pre-menopausal and are not practising an acceptable method of contraception.
19. Treatment with any other investigational agent.
20. Presence of any disease that is likely to shorten life expectancy to < 1 year.
21. Any condition that in the opinion of the investigator would jeopardise the evaluation of efficacy or safety or be associated with poor adherence to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2003-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Adverse events related to amiodarone use and/or atrial fibrillation itself or underlying heart disease

SECONDARY OUTCOMES:
Quality of life
Number of patients with permanent AF at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle C Van Gelder, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Ahmed S, Ranchor AV, Crijns HJ, Van Veldhuisen DJ, Van Gelder IC; CONVERT investigators. Effect of continuous versus episodic amiodarone treatment on quality of life in persistent atrial fibrillation. Europace. 2010 Jun;12(6):785-91. doi: 10.1093/europace/euq049. Epub 2010 Mar 2. PMID 20200016
- [Derived] Ahmed S, Rienstra M, Crijns HJ, Links TP, Wiesfeld AC, Hillege HL, Bosker HA, Lok DJ, Van Veldhuisen DJ, Van Gelder IC; CONVERT Investigators. Continuous vs episodic prophylactic treatment with amiodarone for the prevention of atrial fibrillation: a randomized trial. JAMA. 2008 Oct 15;300(15):1784-92. doi: 10.1001/jama.300.15.1784. PMID 18854540